CLINICAL TRIAL: NCT02357225
Title: Evaluation of Respiratory and Skeletal Muscle Functions in Response to Acetylcholinesterase Inhibitors in Pompe Disease
Brief Title: A Pilot Study of Pyridostigmine in Pompe Disease
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: The drug was ineffective in improving function in Pompe's disease
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB201200154
Record Dates: First submitted 2015-01-23; First posted 2015-02-06 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Pompe Disease
Keywords: Pompe disease; Pyridostigmine
MeSH Terms: conditions — Glycogen Storage Disease Type II | interventions — Pyridostigmine Bromide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acute Dose of Pyridostigmine (Experimental): Subjects will receive an acute administration of pyridostigmine bromide, calculated on their body weight at clinical exam (1 mg/kg, 60mg max starting dose), and will be monitored for 2 hours post administration. Subjects will also receive a pre- and post-administration single-fiber EMG, respiratory tests and strength tests in order to evaluate the function of the neuromuscular junction. All study subjects will be enrolled in this arm.
  Interventions: Drug: Pyridostigmine Bromide
- Prolonged Use of Pyridostigmine (Experimental): This arm will evaluate the impact of pyridostigmine bromide on respiratory and skeletal muscle function during a 90-day administration period. On Days 1 - 7 subjects will receive 0.5mg/kg of the study drug every 4 hours while awake. On Days 8 - 90 subjects will receive 1.0 mg/kg every 4 hours while awake. Quality of life will also be measured with the SF-36 health survey. Data collection will occur at multiple time points (Days 30 and 90) throughout the study. Subjects will also be contacted at least weekly via telephone. All study subjects will be enrolled in this arm.
  Interventions: Drug: Pyridostigmine Bromide

INTERVENTIONS:
Drug: Pyridostigmine Bromide — Pyridostigmine is an acetylcholinesterase inhibitor, which increases the amount of acetylcholine at the neuromuscular junction. It will be taken orally, either as a tablet or as a syrup.
  Other Names: Mestinon

SUMMARY:
Pyridostigmine is an acetylcholinesterase inhibitor, which degrades acetylcholine at the neuromuscular junction. Based on recent studies, pyridostigmine may be an effective adjuvant treatment for people with Pompe disease, as it increases the functional impact of this neurotransmitter.

Hypothesis: the use of pyridostigmine in Pompe disease will improve transmission of acetylcholine across the neuromuscular junction, skeletal muscle function, respiratory function, and quality of life.

DETAILED DESCRIPTION:
Pompe is a rare disease, which occurs in approximately 1 per 40,000 births. It is a progressive and often fatal neuromuscular disorder resulting from mutation in the gene for acid alpha-glucosidase (GAA), an enzyme necessary to degrade glycogen. Accumulation of glycogen in multiple tissues results in cardiac, respiratory and skeletal muscle dysfunction. Enzyme replacement therapy (ERT) is currently the only treatment available, and although it prolongs survival, adjuvant therapies are needed to help alleviate the dire symptoms of Pompe disease.

Recent data has revealed that degradation of the neuromuscular junction (NMJ) occurs in Pompe disease. Acetylcholinesterase inhibitors (AChEI) are substances that inhibit the AChE enzyme from degrading acetylcholine at the NMJ, and thus increase the functional impact of this neurotransmitter. AChEI are established as a beneficial therapy for individuals with primary diseases of the NMJ, such as myasthenia gravis. Recently, administration of an AChEI was demonstrated to improve NMJ pathology in both mice and individuals affected by other congenital myopathies, including autosomal centronuclear myopathies (CNM), X-linked myotubular myopathy (XLMTM) and mutation of tropomyosin 3 (TPM3). Specifically, both NMJ transmission and motor function were improved. These studies demonstrate that AChEI can be beneficial in myopathy associated with NMJ pathology.

In this study, we will study the acute effects of pyridostigmine on neuromuscular transmission, as well as the prolonged effects on respiratory function, skeletal muscle function and quality of life over a 90 day treatment period.

This project focuses on developing an adjuvant treatment to ERT that targets dysfunction at the NMJ. Our ultimate goal is to reduce the deleterious consequences of Pompe disease and improve the overall quality and duration of life in affected individuals.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females between 8 and 60 years of age;
2. Diagnosis of Pompe disease (protein assay, genotyping, and positive clinical signs)
3. No contraindication to pyridostigmine

Exclusion Criteria:

1. Already receive pyridostigmine as part of their normal clinical care at screening
2. Are pregnant - participants will receive a urine pregnancy test at screening
3. Have received acute administration of antibiotic, corticosteroid, or neuromuscular blockade medications within 30 days prior to screening
4. Any other concurrent medical condition which, in the opinion of the study team, would make the subject inappropriate to participate in the assessments

Ages: 8 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Change in skeletal muscle function (6 Minute Walk Test)(QMT) | Baseline, Day 90
  Quantitative muscle testing and the 6 Minute Walk Test will be used to evaluate skeletal muscle function.
Change in respiratory function (maximal inspiratory pressure, maximal expiratory pressure, and vital capacity) | Baseline, Day 90
  Pulmonary function tests, including maximal inspiratory pressure, maximal expiratory pressure, and vital capacity, will be used to evaluate respiratory function
Change in quality of life [short form 36 (SF-36)] | Baseline, Day 90
  The short form 36 health survey (SF-36) will be used to evaluate quality of life
Evaluate the acute effects of pyridostigmine on neuromuscular junction transmission (Single-fiber EMG) | Baseline
  Single-fiber EMG will be performed on the tibialis anterior pre- and 2 hour post-administration of pyridostigmine. MIP and hand grip will also be tested before and after receiving the study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Barry J Byrne, MD, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida Clinical Research Center, Gainesville, Florida, United States

REFERENCES:
- [Background] Byrne BJ, Falk DJ, Pacak CA, Nayak S, Herzog RW, Elder ME, Collins SW, Conlon TJ, Clement N, Cleaver BD, Cloutier DA, Porvasnik SL, Islam S, Elmallah MK, Martin A, Smith BK, Fuller DD, Lawson LA, Mah CS. Pompe disease gene therapy. Hum Mol Genet. 2011 Apr 15;20(R1):R61-8. doi: 10.1093/hmg/ddr174. Epub 2011 Apr 25. PMID 21518733
- [Background] Falk DJ, Todd AG, Lee S, Soustek MS, ElMallah MK, Fuller DD, Notterpek L, Byrne BJ. Peripheral nerve and neuromuscular junction pathology in Pompe disease. Hum Mol Genet. 2015 Feb 1;24(3):625-36. doi: 10.1093/hmg/ddu476. Epub 2014 Sep 12. PMID 25217571
- [Background] Corti M, Smith BK, Falk DJ, Lawson LA, Fuller DD, Subramony SH, Byrne BJ, Christou EA. Altered activation of the tibialis anterior in individuals with Pompe disease: Implications for motor unit dysfunction. Muscle Nerve. 2015 Jun;51(6):877-83. doi: 10.1002/mus.24444. Epub 2015 Apr 24. PMID 25186912
- [Background] Robb SA, Sewry CA, Dowling JJ, Feng L, Cullup T, Lillis S, Abbs S, Lees MM, Laporte J, Manzur AY, Knight RK, Mills KR, Pike MG, Kress W, Beeson D, Jungbluth H, Pitt MC, Muntoni F. Impaired neuromuscular transmission and response to acetylcholinesterase inhibitors in centronuclear myopathies. Neuromuscul Disord. 2011 Jun;21(6):379-86. doi: 10.1016/j.nmd.2011.02.012. Epub 2011 Mar 25. PMID 21440438
- [Background] Maggi L, Mantegazza R. Treatment of myasthenia gravis: focus on pyridostigmine. Clin Drug Investig. 2011 Oct 1;31(10):691-701. doi: 10.2165/11593300-000000000-00000. PMID 21815707